CLINICAL TRIAL: NCT03713528
Title: Can Intraosseous Antibiotics Improve the Results of Irrigation & Debridement and Prosthetic Retention for PJI?
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: American Association of Hip and Knee Surgeons (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9140
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Joint Infection
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: multicenter, single arm, retrospective/prospective clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Other): The treatment group includes any patient with an acute perioperative periprosthetic infection, acute hematogenous infection, or unresectable infection with a gram positive organism sensitive to vancomycin and treated with intraoperative intraosseous vancomycin. Additionally, patients will be treated with at least 4 weeks of IV antibiotics under guidance of an infectious disease specialist, and indefinite antibiotic chronic suppression.
  Interventions: Drug: Intraoperative Intraosseous Vancomycin

INTERVENTIONS:
Drug: Intraoperative Intraosseous Vancomycin — After debridement and irrigation the interventional group will receive intraosseous vancomycin 500mg in 150ml of normal saline. This solution will be prepared by the hospital pharmacy and administered via an EZ-IO intraosseous cannula. 75ccs of the vancomycin solution will be injected as a bolus. Subsequent to this the remaining 75ccs will be placed in the distal femur just proximal to the femoral component evenly split between the medial and lateral femoral condyles in knees.
  Other Names: Vancomycin

SUMMARY:
Purpose of Study: In order to improve upon the variable results seen in irrigation and debridement for periprosthetic infection, we ask if the use of intraosseous regional administration of antibiotics at the time of irrigation and debridement will improve the modest success of standard irrigation and debridement. We will use the existing literature on standard irrigation and debridement procedures to compare with the results of the irrigation and debridement with the use of intraosseous antibiotics.

Impact Question:

How will this study benefit the patient? Currently when an I&D fails, the patient needs to undergo two more major procedures: 1) implant removal and 2) reimplantation of the prosthesis. Any improvement in the results of a standard irrigation and debridement procedure may decrease the number of patients having to go through further extensive procedures to cure their infection.

DETAILED DESCRIPTION:
Type of Study:

This is a multicenter, single arm, retrospective/prospective clinical trial.

Treatment Group:

• The treatment group includes any patient with an acute perioperative infection, an acute hematogenous, or a chronic infection with unresectable components and treated with intraoperative intraosseous vancomycin during a one-stage debridement protocol. Additionally, patients will be treated with at least 4 weeks of IV antibiotics under guidance of an infectious disease specialist, and indefinite antibiotic chronic suppression.

Surgical and Antibiotic Administration Technique:

Initially, all patients will receive standard weight based cefazolin (1 gram for patients < 80kg, 2 grams for patients between 80-120kg, and 3 grams for patients over 120kg) preoperatively. Our protocol for MRSA positive patients is to use cefazolin and vancomycin preoperatively. Because irrigation and debridement in patients with gram positive infections are frequently done urgently before exact organism identification and sensitivities are available it is important to cover the patient broadly with cefazolin and vancomycin initially.

The treatment group will receive post debridement intraosseous vancomycin as described below. In total knee infections a pneumatic tourniquet must be used for the procedure. After entering the knee joint the following process is followed:

1. Fluid is collected in four syringes and placed into two sets of aerobic and anaerobic adult blood culture bottles,
2. Two synovial tissue cultures from different areas of the joint are obtained and sent for culture,
3. If not enough fluid is obtained send an additional tissue culture,
4. Remaining tissue is sent for final pathologic analysis at the end of the case.

After obtaining cultures radical synovial debridement is performed debriding the inner surface of the entire knee capsule including the posterior capsule of the knee. Modular parts will be removed, that is the polyethylene insert for knees.

Debridement and Irrigation Protocol:

After a complete synovectomy is performed along with extraction of modular parts any exposed metallic parts will be scrubbed with a sterile brush soaked in dilute betadine. A 5-step irrigation protocol will then be used for all surgeries:

1. Pulse lavage with 3 liters of normal saline (NS),
2. Lavage with 100 cc's of 3% H202 and 100 cc's of sterile water, a 50/50 solution left in wound for 2 minutes,
3. Lavage 3 liters NS,
4. Lavage with 1 liter of dilute, sterile Betadine (22.5 ml Betadine/liter NS) - left in wound for 3 minutes
5. Pulse lavage with 3 liters of NS

After debridement and irrigation the interventional group will receive intraosseous vancomycin 500mg in 150ml of normal saline. This dose was selected based on the studies of Young (10) and Clarke (11) who used this dose in two high risk groups (revision TKA and high BMI patients) with no significant side effects or red man syndromes. This solution will be prepared by the hospital pharmacy and administered via an EZ-IO intraosseous cannula. In total knees the cannula will be placed in the proximal medial tibia using a starter drill slightly smaller than the diameter of the cannula to ensure a press fit just distal to the tibia implant in the vicinity of the pes anserine tendons. 75ccs of the vancomycin solution will be injected as a bolus. Subsequent to this the remaining 75ccs will be placed in the distal femur just proximal to the femoral component evenly split between the medial and lateral femoral condyles.

After irrigation and debridement the wound will be closed over a betadine soaked lap sponge placed between the components. Contaminated drapes and instruments will be removed and the patient will be re-prepped with new drapes. New instruments will be used to insert the new modular parts. After opening the wound and prior to inserting new modular parts the wound will be irrigated this time with the following regime:

1. Pulse lavage with 3 liters of normal saline (NS),
2. Lavage with 100 cc's of 3% H202 and 100 cc's of sterile water, a 50/50 solution left in wound for 2 minutes,
3. Lavage 1 liters NS,
4. Lavage with 1 liter of dilute, sterile Betadine (22.5 ml Betadine/liter NS) - left in wound for 3 minutes
5. Pulse lavage with 3 liters of NS

After the modular parts are reinserted the wound is closed with monofilament sutures over drains.

Post-operative treatment will be managed by an infectious disease specialist with at least four weeks of intravenous antibiotics followed by indefinite chronic suppression as recommended by the Musculoskeletal Infection Society (Table 1). Baseline creatinine will be obtained preoperatively and on postop days 1 and 2. Infectious disease consultants will monitor peak and trough levels based on the specific antibiotic administered and they will adjust dosage as indicated.

ELIGIBILITY:
Inclusion Criteria (to be completed at time of consent) I. Acute perioperative periprosthetic infection in the first 90 days following primary surgery OR, II. Acute hematogenous infection with symptoms less than four weeks OR, III. Any patient with a chronic periprosthetic knee infection, or a prosthetic knee that is considered unresectable due to the presence of extremely difficult to extract implants such as cones/sleeves/or long cemented or cementless stems and indicated for an irrigation debridement procedure.

IV. Patients indicated for an irrigation debridement procedure of a knee periprosthetic knee joint infection as defined by the inclusion criteria noted above with a gram positive organism susceptible to vancomycin, defined as:

1. A sinus communicating with the prosthesis, OR
2. Two positive cultures obtained from the prosthesis, OR
3. 3 of 5 criteria:

i. Elevated ESR (>30mm/hr) and CRP (>10mg/L) ii. Elevated synovial leukocyte count (>3000 cells/µL) or change of ++ on leukocyte esterase strip iii. Elevated synovial neutrophil percentage (>80%) iv. One positive culture v. Positive histological analysis of periprosthetic tissue (>5 neutrophils per high power field in 5 high power fields x400) We understand that on occasion, irrigation & debridement is performed emergently, therefore enrollment may continue without all laboratory/cultures completed. All inclusion criteria in this situation will be confirmed postoperatively.

V. Any patient >18 years old

Exclusion Criteria I. Surgical wound that cannot be closed. II. Patients with an acute PJI greater than 90 days following primary surgery (using standard implants).

III. Hematogenous infection with symptoms greater than four weeks IV. Know hypersensitivity to Vancomycin V. Major Renal disease defined as creatinine > 2.0 (See previous comments, No Red Man syndrome in 2 subsequent studies on intraosseous vancomycin in revision TKA and High BMI patients respectively (9). Additionally, systemic levels were 8 times lower with intraosseous antibiotics than IV Vancomycin.) VI. Unable to use a tourniquet due to vascular disease VII. Pregnant women VIII. Allergy to antibiotic

Screen Failure (following initial procedure):

IX. Culture negative infections whereby the infecting organism was not identified OR X. Vancomycin-resistant organisms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Infection | 1 year
  The primary outcome measured will be the recurrence of infection by the same organism or reinfection with a new organism as determined by the criteria using the International Consensus Meeting on PJI (1 year follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fehring, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (10):
- United States (10):
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Rush University, Chicago, Illinois
  - University of Nebraska, Omaha, Nebraska
  - New York University - Langone, New York, New York
  - Atrium Mercy Hospital, Charlotte, North Carolina
  - OrthoCarolina Research Institute/OrthoCarolina, Charlotte, North Carolina
  - Novant Health Charlotte Orthopedic Hospital, Charlotte, North Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartman MB, Fehring TK, Jordan L, Norton HJ. Periprosthetic knee sepsis. The role of irrigation and debridement. Clin Orthop Relat Res. 1991 Dec;(273):113-8. PMID 1959257
- [Background] Bradbury T, Fehring TK, Taunton M, Hanssen A, Azzam K, Parvizi J, Odum SM. The fate of acute methicillin-resistant Staphylococcus aureus periprosthetic knee infections treated by open debridement and retention of components. J Arthroplasty. 2009 Sep;24(6 Suppl):101-4. doi: 10.1016/j.arth.2009.04.028. Epub 2009 Jun 24. PMID 19553077
- [Background] Fehring TK, Odum SM, Berend KR, Jiranek WA, Parvizi J, Bozic KJ, Della Valle CJ, Gioe TJ. Failure of irrigation and debridement for early postoperative periprosthetic infection. Clin Orthop Relat Res. 2013 Jan;471(1):250-7. doi: 10.1007/s11999-012-2373-9. PMID 22552768
- [Background] Bryan AJ, Abdel MP, Sanders TL, Fitzgerald SF, Hanssen AD, Berry DJ. Irrigation and Debridement with Component Retention for Acute Infection After Hip Arthroplasty: Improved Results with Contemporary Management. J Bone Joint Surg Am. 2017 Dec 6;99(23):2011-2018. doi: 10.2106/JBJS.16.01103. PMID 29206791
- [Background] Urish KL, Bullock AG, Kreger AM, Shah NB, Jeong K, Rothenberger SD; Infected Implant Consortium. A Multicenter Study of Irrigation and Debridement in Total Knee Arthroplasty Periprosthetic Joint Infection: Treatment Failure Is High. J Arthroplasty. 2018 Apr;33(4):1154-1159. doi: 10.1016/j.arth.2017.11.029. Epub 2017 Nov 21. PMID 29221840
- [Background] Young SW, Zhang M, Freeman JT, Vince KG, Coleman B. Higher cefazolin concentrations with intraosseous regional prophylaxis in TKA. Clin Orthop Relat Res. 2013 Jan;471(1):244-9. doi: 10.1007/s11999-012-2469-2. PMID 22773397
- [Background] Young SW, Zhang M, Freeman JT, Mutu-Grigg J, Pavlou P, Moore GA. The Mark Coventry Award: Higher tissue concentrations of vancomycin with low-dose intraosseous regional versus systemic prophylaxis in TKA: a randomized trial. Clin Orthop Relat Res. 2014 Jan;472(1):57-65. doi: 10.1007/s11999-013-3038-z. PMID 23666589
- [Background] Young SW, Roberts T, Johnson S, Dalton JP, Coleman B, Wiles S. Regional Intraosseous Administration of Prophylactic Antibiotics is More Effective Than Systemic Administration in a Mouse Model of TKA. Clin Orthop Relat Res. 2015 Nov;473(11):3573-84. doi: 10.1007/s11999-015-4464-x. Epub 2015 Jul 30. PMID 26224291
- [Background] Young SW, Zhang M, Moore GA, Pitto RP, Clarke HD, Spangehl MJ. The John N. Insall Award: Higher Tissue Concentrations of Vancomycin Achieved With Intraosseous Regional Prophylaxis in Revision TKA: A Randomized Controlled Trial. Clin Orthop Relat Res. 2018 Jan;476(1):66-74. doi: 10.1007/s11999.0000000000000013. PMID 29529618
- [Background] Chin SJ, Moore GA, Zhang M, Clarke HD, Spangehl MJ, Young SW. The AAHKS Clinical Research Award: Intraosseous Regional Prophylaxis Provides Higher Tissue Concentrations in High BMI Patients in Total Knee Arthroplasty: A Randomized Trial. J Arthroplasty. 2018 Jul;33(7S):S13-S18. doi: 10.1016/j.arth.2018.03.013. Epub 2018 Mar 15. PMID 29655497
- [Background] Lichstein P, Gehrke T, Lombardi A, Romano C, Stockley I, Babis G, Bialecki J, Bucsi L, Cai X, Cao L, de Beaubien B, Erhardt J, Goodman S, Jiranek W, Keogh P, Lewallen D, Manner P, Marczynski W, Mason JB, Mulhall K, Paprosky W, Patel P, Piccaluga F, Polkowski G, Pulido L, Stockley I, Suarez J, Thorey F, Tikhilov R, Velazquez JD, Winkler H. One-stage vs two-stage exchange. J Arthroplasty. 2014 Feb;29(2 Suppl):108-11. doi: 10.1016/j.arth.2013.09.048. Epub 2013 Oct 1. No abstract available. PMID 24360339